CLINICAL TRIAL: NCT03980015
Title: Inflammatory Responses in Borrelia Afzelii Culture Positive Patients With Early Disseminated or Early Localized Lyme Borreliosis
Brief Title: Inflammatory Responses in Solitary and Multiple Erythema Migrans
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: University of Ljubljana School of Medicine, Slovenia (Other)
Responsible Party: Principal Investigator, Daša Stupica, Prinicipal Investigator, University Medical Centre Ljubljana
Other Study IDs: MEM vs EM cyto
Record Dates: First submitted 2019-06-05; First posted 2019-06-10 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Erythema Migrans
MeSH Terms: conditions — Glossitis, Benign Migratory

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- erythema migrans: patients with erythema migrans
  Interventions: Other: antibiotic treatment

INTERVENTIONS:
Other: antibiotic treatment — Patients were treated with: ceftriaxone intravenously 2 g OD for 14 days or doxycycline orally 100 mg bid for 10 to 14 days or cefuroxime axetil orally 500 mg bid for 14 days or amoxicillin orally 500 mg tid for 14 days

SUMMARY:
The investigators will evaluate differences in host immune responses (levels of cytokines and chemokines, representative of innate, Th1, and Th17 immune responses) in acute sera from adult patients with solitary or multiple erythema migrans.

ELIGIBILITY:
Inclusion Criteria:

* erythema migrans in patients > 18 years
* Borrelia afzelii isolated from skin

Exclusion Criteria:

* pregnancy or immunocompromising conditions
* taking antibiotic with antiborrelial activity within 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with erythema migrans
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
inflammatory proteins in erythema migrans patients | at enrollment
  The inflammatory immune profiles will be assessed using Luminex to measure the expression of cytokines and chemokines representative of innate and adaptive TH1, TH2, TH17, and B cell responses in serum of patients at enrollment (during active infection).

CONTACTS AND LOCATIONS:
Overall Officials: Daša Stupica, MD PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided